CLINICAL TRIAL: NCT05866211
Title: Associated Factors for Impaired Lung Function in Post-COVID Nursing Home Residents
Brief Title: Lung Function in Post-COVID-19 Nursing Home Residents
Status: Completed | Type: Observational
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: Catalan Board of Physiotherapists (Unknown)
Responsible Party: Sponsor
Other Study IDs: LUNGFUNCTIONCFCR101
Record Dates: First submitted 2023-05-11; First posted 2023-05-19 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2023-05

CONDITIONS: Post-COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case: Individuals with impaired lung function, according to spirometry results (FVC ≤ LLN and FEV1/FVC ≥ LLN).
  Interventions: Other: Previous exposure to SARS-CoV-2
- Control: Individuals with normal lung function
  Interventions: Other: Previous exposure to SARS-CoV-2

INTERVENTIONS:
Other: Previous exposure to SARS-CoV-2 — This is an observational study in which no intervention will be applied.

SUMMARY:
The coronavirus disease 2019 (COVID-19) took a toll in institutionalised older adults, who represent a vulnerable population in European countries.

The aim of this study is to identify the predictive factors that worsens lung function in post-COVID nursing home (NH) residents.

This is a multicenter case-control study in nursing homes of Osona (Catalonia), where individuals with worsened (cases) and normal (controls) lung function will be studied. The inclusion criteria are: female and male from 65 to 95 years old, preserved cognitive capacity and positive diagnosis of COVID-19 at least 3 months prior.

We will assess sociodemographic variables, lung function [spirometry], fatigue [Chalder Fatigue Scale], frailty [Clinical Frailty Scale], and activities of daily living (ADL) [modified Barthel index].

ELIGIBILITY:
Inclusion Criteria:

* male and female
* preserved cognitive function
* previous positive diagnosis of COVID-19 at a minimum of 3 months to the day of data collection
* individuals living permanently in a nursing home

Exclusion Criteria:

* individuals in coma or palliative care
* any contraindication to perform spirometry (severe hypertension, myocardial infarction in the past week, non compensated heart failure, etc).

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The population will be institutionalised older adults previously infected with SARS-CoV-2, either symptomatic or asymptomatic.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Lung function | Through study completion, an average of 1 year
  Lung function will be assessed by spirometry.

SECONDARY OUTCOMES:
Sociodemographic variables | Through study completion, an average of 1 year
  Sociodemographic variables (age, gender, length of institutionalization) will be collected through an interview.
Anthropometric variables | Through study completion, an average of 1 year
  Anthropometric variables (weight and height) will be collected by means of a scale and a measuring tape, respectively.
Health variables | Through study completion, an average of 1 year
  Health variables (history of comorbidities) will be collected directly in the medical records of each participant.
COVID-19 variables | Through study completion, an average of 1 year
  The following variables related to COVID-19 will be collected from the medical records of each participant: diagnostic tests (PCR and serological test), suspicious case (symptoms of cough, fever, difficulty breathing, etc.), previous hospitalization for COVID-19 (yes/no, duration), use of mechanical ventilation during hospitalization (yes/no, duration) and vaccination (yes/no, type).
Fatigue | Through study completion, an average of 1 year
  Fatigue levels will be collected using the Chalder Fatigue Scale (CFQ-11)
Frailty | Through study completion, an average of 1 year
  Frailty levels will be assessed using the Clinical Frailty Scale (CFS).
Dependency levels | Through study completion, an average of 1 year
  Dependency levels will be assessed using the Barthel modified index.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences and Welfare, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Research data cannot be shared due to ethical issues regarding patients' privacy according to the Research Ethics Committee of the University of Vic - Central University of Catalonia (Spain). Only the study results may be shared.